CLINICAL TRIAL: NCT02170090
Title: Adjuvant Chemotherapy With Gemcitabine and Cisplatin Compared to Standard of Care After Curative Intent Resection of Cholangiocarcinoma and Muscle Invasive Gall Bladder Carcinoma (ACTICCA-1 Trial)
Brief Title: Adjuvant Chemotherapy With Gemcitabine and Cisplatin Compared to Standard of Care After Curative Intent Resection of Biliary Tract Cancer
Acronym: ACTICCA-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Cancer Research UK (Other); Australasian Gastro-Intestinal Trials Group (Network); Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTICCA-1; 2024-517340-61-00 (EU CTIS Number); ACTRN12615001283561 (Registry Identifier: ANZCTR (clinical trial registry))
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cholangiocarcinoma; Gall Bladder Carcinoma
Keywords: adjuvant chemotherapy; cholangiocarcinoma; muscle invasive gall bladder carcinoma; translational research; multidisciplinary; AIO, DGAV, DGVS
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Gemcitabine; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine plus Cisplatin (Experimental): Chemotherapy will be administered on days 1 and 8 every 3 weeks, Cisplatin (25 mg per square meter of body-surface area) and Gemcitabine (1000 mg per square meter) for 24 weeks (8 cycles)
  and Observation
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- Capecitabine (Active Comparator): Capecitabine will be administered from day 1 to 14 every 3 weeks (1250 mg per square meter of body-surface area, twice daily) for 24 weeks (8 cycles)
  and Observation
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m2
  Arms: Gemcitabine plus Cisplatin
Drug: Cisplatin — Cisplatin 25mg/m2
  Arms: Gemcitabine plus Cisplatin
Drug: Capecitabine — Capecitabine 1250mg/m2
  Arms: Capecitabine

SUMMARY:
This is a multicenter, prospective, randomized, controlled phase III trial designed to assess the clinical performance of gemcitabine with cisplatin and observation vs. standard of care (observation alone in stage 1 and capecitabine and observation in stage 2) in patients after curative intent resection of BTC.

DETAILED DESCRIPTION:
The ACTICCA-1 investigator initiated trial is funded by the Deutsche Krebshilfe (grant number 70110215, 70112047). With respect to data obtained in the ABC-02 trial, the combination of cisplatin and gemcitabine for 24 weeks as investigational treatment was selected. Based on adjuvant trials in pancreatic cancer (e.g. ESPAC IV) with a comparable postoperative recovery time, inclusion of patients within a maximum interval of 16 weeks between surgery and start of CTx was chosen. Gemcitabine and cisplatin has a relevantly higher cumulative dose of gemcitabine 18 vs. 12 applications and may thus be of increased efficacy compared to the gemcitabine/oxaliplatin regimen applied in the PRODIGE 12 trial.

Based on the data of the BILCAP trial showing an improvement in median overall survival for capecitabine compared to observation alone presented at the annual meeting of the American Society of Clinical Oncology on June 4th 2017 in Chicago by the British BILCAP trial group, capecitabine has evolved as the new standard of care after curative intent resection of biliary tract cancer.

Based on these data the comparative efficacy of gemcitabine/cisplatin and capecitabine had to be established.

Therefore, the ACTICCA trial was amended to compare gemcitabine and cisplatin to the newly established standard regimen in the adjuvant setting capecitabine, aiming for superiority of the combination regimen vs. the oral monotherapy This was based on the BILCAP protocol, applying the similar dosing, assessments and dose modifications as in BILCAP, including dose calculation and patient diary.

As data of recent trials like the French PRODIGE 12/ACCORD 18 trial have clearly shown that in terms of efficacy of an adjuvant chemotherapy there is no difference between cholangiocarcinoma and gall bladder carcinoma, these two subtypes are pooled and location was added as an stratification factor.

Randomization will be 1:1 with adjuvant CTx for 24 weeks and imaging every 12 weeks in the experimental arm and standard of care (capecitabine) and observation in the control arm.

The primary endpoint is DFS and secondary endpoints include recurrence free survival, OS, safety and tolerability of adjuvant CTx, quality of life, and patterns of disease recurrence.

ELIGIBILITY:
All enrolled patients will postoperatively be assessed for eligibility for the treatment phase. Additionally patients not previously enrolled into the trial for whatever reason (e.g. incidental finding during surgery) will be evaluated for eligibility.

* Histologically confirmed adenocarcinoma of biliary tract (intrahepatic, hilar or extrahepatic cholangiocarcinoma or muscle invasive gallbladder carcinoma) after radical surgical therapy with macroscopically complete resection (mixed tumor entities (HCC/CCA) are excluded)
* Macroscopically complete resection (R0/1) within 6 (-16) weeks before scheduled start of chemotherapy
* ECOG 0-1
* Age ≥18 years
* Adequate hematologic function
* Adequate liver function
* Adequate renal function
* No active uncontrolled infection, except chronic viral hepatitis under antiviral therapy
* No concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to randomization
* Negative serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women <1 year after the onset of menopause (Note: a negative test has to be reconfirmed by a urine test, should the 7-day window be exceeded)

Criteria for initial study enrolment

* Written informed consent
* No prior chemotherapy for cholangiocarcinoma
* No previous malignancy within 3 years or concomitant malignancy, except: non-melanomatous skin cancer or adequately treated in situ cervical cancer
* No severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction in the last 3 months, significant arrhythmia)
* Absence of psychiatric disorder precluding understanding of information of trial related topics and giving informed consent
* No serious underlying medical conditions (judged by the investigator), that could impair the ability of the patient to participate in the trial
* Fertile women (< 1 year after last menstruation) and procreative men willing and able to use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)
* No pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2014-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Disease free survival rate at 24 months (DFSR@24)
  DFS

SECONDARY OUTCOMES:
Disease free survival rate at 24 months (DFSR@24) | 24 months
  DSFR
Recurrence free survival | 24 months
  RFS
Overall survival | 84 months
  OS
Safety and tolerability (assessed by the rate of patients with adverse events according to NCI CTC AE v4.03) | 24 months
Quality of life | 48 months
  QOL
Function of biliodigestive anastomosis (in terms of surgical revision, requirement for PTCD) | 48 months
Rate and severity of biliary tract infections | 48 months
Patterns of disease recurrence | 48 months
locoregional control (assessed by the rate of patients with hepatic or locoregional recurrence) | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Wege, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (67):
- Australia (12):
  - Bankstown Hospital, Bankstown, New South Wales
  - Nepean Hospital Cancer Care, Kingswood, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Fiona Stanley Hospital Perth, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St. John of God, Subiaco, Western Australia
- Kaiser-Franz-Josef Hospital, Vienna, Austria
- Vejle Hospital, Vejle, Denmark
- Germany (19):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - University Medical Center Aachen, Aachen
  - Charite Berlin, Berlin
  - University Medical Center Carl Gustav Carus, Dresden
  - University Medical Center Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - University of Frankfurt, Frankfurt
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University of Hannover, Hanover
  - University of Heidelberg, Heidelberg
  - University of Saarland, Homburg
  - University Medical Center Jena, Jena
  - Johannes Gutenberg University of Mainz, Mainz
  - University of Mannheim, Mannheim
  - University of Munich Grosshadern, Munich
  - University of Regensburg, Regensburg
  - University Medical Center Tuebingen, Tübingen
  - University of Ulm, Ulm
  - University Medical Center, Würzburg
- Italy (5):
  - Istituto Oncologico Veneto IRCCS, Padua, Padova
  - Azienda Ospedaliero Medica 2 Universitaria, Pisa, Pisa
  - Fondazione Policlinico Gemelli, Roma, Rome, Rome
  - Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Auckland Hospital, Auckland, New Zealand
- United Kingdom (24):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital Cambridge, Cambridge
  - Velindre Hospital Cardiff, Cardiff
  - Western General Hospital Edinburgh, Edinburgh
  - Beatson West of Scotland Cancer Centre Glasgow, Glasgow
  - James Paget University Hospitals, Great Yarmouth
  - Royal Surrey County Hospital Guildford, Guildford
  - Princess Alexandra Hospital, Harlow
  - Huddersfield Royal Infirmary, Huddersfield
  - Guy's and St Thomas's Hospital London, London
  - Hammersmith Hospital London, London
  - Royal Free Hospital London, London
  - University College London Hospital, London
  - Maidstone Hospital, Maidstone
  - Christie Hospital Manchester, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital Oxford, Oxford
  - Derriford Hospital Plymouth, Plymouth
  - Weston Park Hospital Sheffield, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stein A, Arnold D, Bridgewater J, Goldstein D, Jensen LH, Klumpen HJ, Lohse AW, Nashan B, Primrose J, Schrum S, Shannon J, Vettorazzi E, Wege H. Adjuvant chemotherapy with gemcitabine and cisplatin compared to observation after curative intent resection of cholangiocarcinoma and muscle invasive gallbladder carcinoma (ACTICCA-1 trial) - a randomized, multidisciplinary, multinational phase III trial. BMC Cancer. 2015 Jul 31;15:564. doi: 10.1186/s12885-015-1498-0. PMID 26228433